CLINICAL TRIAL: NCT04598256
Title: Evaluation of Children Who Were Underwent Endoscopic Procedures in the Normalization Process of Covid-19 Pandemic
Brief Title: Endoscopic Procedures of Children in the Normalization Process of Covid-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Tepecik Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Prof. masallah Baran, professor, Tepecik Training and Research Hospital
Other Study IDs: TepecikTRH1
Record Dates: First submitted 2020-10-21; First posted 2020-10-22 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: endoscopy; colonoscopy; children; Covid -19 pandemic
MeSH Terms: conditions — COVID-19 | interventions — Endoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children who underwent endoscopic procedures: * Children between the ages of 1-18 who were underwent endoscopic procedures
  * Patients who can be questioned about COVID-19 infection before and on the 7th and 14th days after the procedure
  * Patients who volunteered to study
  Interventions: Procedure: Endoscopic procedure

INTERVENTIONS:
Procedure: Endoscopic procedure — Esophagogastroscopy and colonoscopy

SUMMARY:
Endoscopic methods are frequently used in the diagnosis of gastrointestinal system pathologies in children.

DETAILED DESCRIPTION:
Endoscopic methods are frequently used in the diagnosis of gastrointestinal system pathologies in children. In the investigators' center, which is a pandemic hospital, only emergency endoscopic procedures were performed during the pandemic period, while emergency and elective endoscopic procedures are performed in accordance with the recommendations of the Ministry of Health during the normalization process. Staff and patients in endoscopy units are at risk for COVID-19 infection by inhalation of airborne droplets, conjunctival contact, and potential fecal-oral contamination. In order to reduce the risk of contamination, according to the recommendations of the European Gastrointestinal Endoscopy Association (ESGE); proper cleaning of endoscopic devices, non-reuse of disposable devices, cleaning the endoscopy hall with a disinfectant solution, use of gowns FFP2 / 3 masks and jewelry during the procedure, handwashing with soap and hand disinfection is recommended before and after each procedure. In addition, it is recommended that patients who have undergone endoscopic procedures should be followed up or communicated on days 7 and 14 in terms of the development of COVID-19 infection.

It is recommended that patients should be questioned in terms of COVID-19 infection before endoscopy, but rapid antigen testing and serology are not routinely recommended. Molecular diagnosis (PCR, amplification) tests are recommended for patients at risk for COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 1-18 who will undergo endoscopic procedures
* Patients who can be questioned about COVID-19 infection before and on the 7th and 14th days after the procedure
* Patients who volunteered to study

Exclusion Criteria:

* Under 1 year and over 18 years of age
* Patients who could not be questioned about COVID-19 infection before the procedure and on the 7th and 14th days after the procedure
* Patients who not volunteered to study

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients aged 1 to 18 years who underwent emergency or elective endoscopic procedures will be included in the study. Demographic characteristics of the patients, indication of the procedure, date, place of operation, procedure performed and endoscopic diagnosis will be noted. Before and on the 7th and 14th days after the procedure, patients will be contacted and the symptoms and clinical findings in terms of COVID-19 infection will be questioned and noted. The results of complete blood count, CRP, coagulation profile, COVID-19 PCR, chest radiography and thorax computed tomography will be recorded if it was performed on the patient.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
The number of participiants who was infected with Covid-19. normalization process of Covid-19 pandemic | 14 days
  The number of participiants who had Covid-19 infection after the endoscopic procedures.
The time of seen covid 19 infection after the endoscopic procedures in participiants. | 14 days
  The developed time of covid 19 infection after the endoscopic procedures in participiants.
The characteristics of patients with Covid-19 infection. | 14 days
  The characteristics of patients with Covid-19 infection after the endoscopic procedures in participiants.

CONTACTS AND LOCATIONS:
Overall Officials: BETÜL AKSOY, MD, Study Chair — Yes; YELİZ ÇAĞAN APPAK, MD, Study Chair — Yes; DİLEK YILMAZ ÇİFTDOĞAN, PROFESSOR, Study Chair — Yes; MAŞALLAH BARAN, PROFESSOR, Principal Investigator — Yes; ŞENAY ONBAŞI KARABAĞ, MD, Study Chair — Yes
Locations (1):
- Tepecik Trh, Izmir, İ̇zmi̇r, Turkey (Türkiye)

REFERENCES:
- [Background] Gralnek IM, Hassan C, Beilenhoff U, Antonelli G, Ebigbo A, Pellise M, Arvanitakis M, Bhandari P, Bisschops R, Van Hooft JE, Kaminski MF, Triantafyllou K, Webster G, Pohl H, Dunkley I, Fehrke B, Gazic M, Gjergek T, Maasen S, Waagenes W, de Pater M, Ponchon T, Siersema PD, Messmann H, Dinis-Ribeiro M. ESGE and ESGENA Position Statement on gastrointestinal endoscopy and the COVID-19 pandemic. Endoscopy. 2020 Jun;52(6):483-490. doi: 10.1055/a-1155-6229. Epub 2020 Apr 17. PMID 32303090
- [Background] Gralnek IM, Hassan C, Beilenhoff U, Antonelli G, Ebigbo A, Pellise M, Arvanitakis M, Bhandari P, Bisschops R, Van Hooft JE, Kaminski MF, Triantafyllou K, Webster G, Voiosu AM, Pohl H, Dunkley I, Fehrke B, Gazic M, Gjergek T, Maasen S, Waagenes W, de Pater M, Ponchon T, Siersema PD, Messmann H, Dinis-Ribeiro M. ESGE and ESGENA Position Statement on gastrointestinal endoscopy and COVID-19: An update on guidance during the post-lockdown phase and selected results from a membership survey. Endoscopy. 2020 Oct;52(10):891-898. doi: 10.1055/a-1213-5761. Epub 2020 Jul 14. No abstract available. PMID 32643767
- See also: PubMed ID: 32303090 — https://www.esge.com/esge-and-esgena-position-statement-on-gastrointestinal-endoscopy-and-the-covid-19-pandemic/
- See also: PubMed ID: 32643767 — https://www.esge.com/update-on-esge-and-esgena-position-statement-on-gastrointestinal-endoscopy-and-covid-19/